CLINICAL TRIAL: NCT02616146
Title: A Phase 3, Randomized, Active-Comparator Controlled Clinical Trial to Study the Contraceptive Efficacy and Safety of the MK-8342B (Etonogestrel + 17β-Estradiol) Vaginal Ring and the Levonorgestrel-Ethinyl Estradiol (LNG-EE) 150/30 μg Combined Oral Contraceptive (COC) in Healthy Women 18 Years of Age and Older, at Risk for Pregnancy.
Brief Title: Efficacy and Safety of Etonogestrel + 17β-Estradiol Vaginal Ring and Levonorgestrel-Ethinyl Estradiol Combined Oral Contraceptive in Adult Women at Risk for Pregnancy (MK-8342B-062)
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Study terminated by Sponsor as a result of a business decision to discontinue the development program for MK-8342B for reasons unrelated to safety or efficacy.
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 8342B-062; 2014-002208-26 (EudraCT Number); MK-1029-006 (Other: Merck Protocol Number)
Record Dates: First submitted 2015-11-24; First posted 2015-11-26 (Estimated); Results first posted 2019-01-18 (Actual); Last update posted 2024-05-17 (Actual); Status verified 2022-02

CONDITIONS: Contraception
MeSH Terms: interventions — Contraceptive Devices, Female; etonogestrel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ENG-E2 125 μg/300 μg (Experimental): Participants will receive up to 13 cycles of ENG-E2 125 μg/300 μg. Each cycle will consist of 21 days of vaginal ring use followed by 7 vaginal ring-free days.
  Interventions: Drug: ENG-E2 125 μg/300 μg vaginal ring
- LNG-EE 150 μg/30 μg (Active Comparator): Participants will receive up to 13 cycles of LNG-EE 150 μg/30 μg. Each cycle will consist of one tablet per day for 21 days, followed a 7-day tablet-free interval.
  Interventions: Drug: LNG-EE 150 μg/30 μg COC

INTERVENTIONS:
Drug: ENG-E2 125 μg/300 μg vaginal ring — Up to 13 cycles of ENG-E2 125 μg/300 μg administered intravaginally, each cycle consisting of 21 days of vaginal ring use followed by 7 vaginal ring-free days.
  Other Names: Etonogestrel + 17β-Estradiol Vaginal Ring
  Arms: ENG-E2 125 μg/300 μg
Drug: LNG-EE 150 μg/30 μg COC — Up to 13 cycles of LNG-EE 150 μg/30 μg administered orally, each cycle consisting of one tablet per day for 21 days, followed a 7-day tablet-free interval.
  Other Names: Levonorgestrel-Ethinyl Estradiol COC
  Arms: LNG-EE 150 μg/30 μg

SUMMARY:
The purpose of this study is to assess the contraceptive efficacy of the etonogestrel + 17β-estradiol (ENG-E2) vaginal ring in women between 18 and 35 years of age based on the number of in-treatment pregnancies as expressed by the Pearl Index (PI). The study will also assess the safety and tolerability of ENG-E2 vaginal ring. The levonorgestrel-ethinyl estradiol (LNG-EE) 150/30 μg combined oral contraceptive (COC) will be used as the active comparator.

ELIGIBILITY:
Inclusion Criteria:

* Premenopausal female at risk for pregnancy and seeking contraception.
* Willing to use a hormonal contraceptive vaginal ring for up to 13 treatment cycles, and not intending to use any other form of contraception.
* Body mass index (BMI) of ≥18 and <38 kg/m^2.
* In good physical and mental health, based upon the medical judgment of the investigator.
* Willing to adhere to use of vaginal ring and all required trial procedures.

Exclusion Criteria:

* Cardiovascular risks and disorders, including history of venous thromboembolic [VTE] events, arterial thrombotic or thromboembolic [ATE] events, transient ischemic attack, angina pectoris, or claudication; at higher risk of VTE events due to recent prolonged immobilization, plans for surgery requiring prolonged immobilization, or a hereditary or acquired predisposition or elevated risk for venous or arterial thrombosis; currently smoking or uses tobacco/nicotine containing products and is ≥35 years of age; uncontrolled or severe hypertension; history of severe dyslipoproteinemia; <35 years of age with a history of migraine with aura or focal neurological symptoms or ≥35 years of age with a history of migraines with or without aura or focal neurologic symptoms; diabetes mellitus with end-organ involvement or >20 years duration; multiple cardiovascular risk factors such as ≥35 years of age, obesity, inadequately controlled hypertension, use of tobacco/ nicotine products, or inadequately controlled diabetes.
* Gastrointestinal disorders, including history of pancreatitis associated with severe hypertriglyceridemia; clinically significant liver disease, including active viral hepatitis or cirrhosis; history of malabsorptive bariatric surgery.
* Other medical disorders, including history of malignancy ≤5 years prior to signing informed consent except for adequately treated basal cell or squamous cell skin cancer or in situ cervical cancer; any disease that may worsen under hormonal treatment such as disturbances in bile flow, systemic lupus erythematosus, pemphigoid gestationis or idiopathic icterus during previous pregnancy, middle-ear deafness, Sydenham chorea, or porphyria; known allergy/sensitivity or contraindication to the investigational products or their excipients; history of drug or alcohol abuse or dependence.
* Recent, current, or suspected pregnancy; or has not had at least 2 menstrual cycles or has not completed two 28-day cycles of a hormonal contraceptive following a recent pregnancy; or is breastfeeding.
* Gynecologic conditions: has gonorrhea, chlamydia, or trichomonas or symptomatic vaginitis/cervicitis; has abnormal cervical Pap test or positive high-risk human papillomavirus (HPV) test at screening or documented within 3 years of screening; currently using an intrauterine device/intrauterine system (IUD/IUS) or contraceptive implant; within past 6 months has had undiagnosed (unexplained) abnormal vaginal bleeding or any abnormal vaginal bleeding expected to recur during trial; has stage 4 pelvic organ prolapse (1 cm beyond introitus) or lesser degrees of prolapse with history of difficulty retaining tampons, vaginal rings, or other products within vagina.
* Has used investigational drug and/or participated in other clinical trial within past 8 weeks.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2016 (Actual)
Dates: Start 2015-12-01 (Actual); Primary Completion 2016-10-06 (Actual); Study Completion 2016-10-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (14):
- MSD Osterreich GmbH, Vienna, Austria
- Merck Sharp & Dohme, San José, Costa Rica
- Merck Sharp & Dohme, Glostrup Municipality, Denmark
- MSD Finland Oy, Espoo, Finland
- Merck Sharp & Dohme GmbH, Haar, Germany
- MSD Pharma Hungary Kft., Budapest, Hungary
- MSD Italia S.r.l., Rome, Italy
- MSD, Mexico City, Mexico
- Merck Sharp & Dohme BV, Haarlem, Netherlands
- MSD Norge A/S, Drammen, Norway
- Merck Sharp & Dohme, Peru S.R.L., Lima, Peru
- MSD Polska Sp. Z o.o., Warsaw, Poland
- MSD (Pty) LTD South Africa, Midrand, South Africa
- MSD Sweden, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Note: One participant less than 18 years of age was inadvertently randomized and received study medication. She was discontinued from the study due to the major protocol violation.
Groups:
- ENG-E2 125 μg/300 μg: Participants were to receive up to 13 cycles of etonogestrel + 17β-estradiol (ENG-E2) 125 μg/300 μg. Each cycle was to consist of 21 days of vaginal ring use followed by 7 vaginal ring-free days.
- LNG-EE 150 μg/30 μg: Participants were to receive up to 13 cycles of levonorgestrel-ethinyl estradiol (LNG-EE) 150 μg/30 μg. Each cycle was to consist of one tablet per day for 21 days, followed a 7-day tablet-free interval.
Period: Overall Study
Arm/Group | ENG-E2 125 μg/300 μg | LNG-EE 150 μg/30 μg
Started | 1512 | 504
Completed | 0 (Due to termination of study, ENG-E2 reporting group received only up to 10 cycles of treatment.) | 0 (Due to termination of study, LNG-EE reporting group received only up to 9 cycles of treatment.)
Not Completed | 1512 | 504
Not completed — Adverse Event | 64 | 24
Not completed — Lost to Follow-up | 23 | 13
Not completed — Non-compliance with study protocol | 2 | 0
Not completed — Non-compliance with study drug | 4 | 2
Not completed — Pregnancy | 2 | 2
Not completed — Pregnancy wish | 3 | 0
Not completed — Protocol Violation | 6 | 3
Not completed — Study terminated by sponsor | 1372 | 432
Not completed — Participant moved | 4 | 3
Not completed — Withdrawal by Subject | 30 | 24
Not completed — Physician Decision | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- ENG-E2 125 μg/300 μg: Participants were to receive up to 13 cycles of ENG-E2 125 μg/300 μg. Each cycle was to consist of 21 days of vaginal ring use followed by 7 vaginal ring-free days.
- LNG-EE 150 μg/30 μg: Participants were to receive up to 13 cycles of LNG-EE 150 μg/30 μg. Each cycle was to consist of one tablet per day for 21 days, followed a 7-day tablet-free interval.
- Total: Total of all reporting groups
Arm/Group | ENG-E2 125 μg/300 μg | LNG-EE 150 μg/30 μg | Total
Number analyzed (Participants) | 1512 | 504 | 2016
Age, Continuous [Mean (Standard Deviation); unit: Years] | 27.5 (6.3) | 27.5 (6.3) | 27.5 (6.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1512 | 504 | 2016
  Male | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of In-Treatment Pregnancies Per 100 Woman-Years of Exposure in Participants 18-35 Years of Age (Pearl Index)
Description: The Primary Efficacy Outcome Measure for this study was contraceptive efficacy, or the prevention of in-treatment pregnancy. The total incidence of in-treatment pregnancies was expressed as the Pearl Index, which is defined as the number of in-treatment pregnancies per 100 woman-years of exposure (one woman-year defined as a period of 365.25 days). NOTE: Due to early termination of this study, the ENG-E2 reporting group received only up to 10 cycles of treatment, and the LNG-EE reporting group received only up to 9 cycles of treatment.
Time Frame: Up to 1 year (13 28-day cycles)
Population: restricted Full Analysis Set (rFAS) population, defined as the population of women with at least one "at risk" treatment cycle without documented use of hormonal or nonhormonal backup contraception during the cycle, or participants with a treatment cycle (at risk or not) in which a pregnancy has occurred.
Measure: Number; unit: Pregnancies per 100 woman years
Arm/Group | ENG-E2 125 μg/300 μg | LNG-EE 150 μg/30 μg
Number analyzed (Participants) | 1266 | 404
Pregnancies per 100 woman years | 1.54 | 2.93

2. Primary Outcome: Number of Participants Who Experienced an Adverse Event (AE)
Description: An AE is any untoward medical occurrence in a participant administered a pharmaceutical product and which does not necessarily have to have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of a medicinal product or protocol-specified procedure, whether or not considered related to the medicinal product or protocol specified procedure. Any worsening (i.e., any clinically significant adverse change in frequency and/or intensity) of a preexisting condition that is temporally associated with the use of the Sponsor's product, is also an AE. NOTE: Due to early termination of this study, the ENG-E2 reporting group received only up to 10 cycles of treatment, and the LNG-EE reporting group received only up to 9 cycles of treatment.
Time Frame: Up to 1 year
Population: This primary endpoint was based on all randomized participants in whom at least one vaginal ring was inserted or one comparator tablet was ingested.
Measure: Count of Participants; unit: Participants
Arm/Group | ENG-E2 125 μg/300 μg | LNG-EE 150 μg/30 μg
Number analyzed (Participants) | 1504 | 492
Participants | 530 | 140

3. Primary Outcome: Number of Participants Who Discontinued Treatment Due to an AE
Description: as for outcome 2
Time Frame: Up to 1 year
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | ENG-E2 125 μg/300 μg | LNG-EE 150 μg/30 μg
Number analyzed (Participants) | 1504 | 492
Participants | 61 | 23

4. Secondary Outcome: Number of Participants With Breakthrough Bleeding/Spotting (BTB-S), by Cycle
Description: BTB-S was considered any bleeding/spotting that occurred during expected non-bleeding interval that was neither early nor continued withdrawal bleeding. BTB-S was classified as follows: Bleeding = any bloody vaginal discharge that required one or more sanitary pads or tampons per day; Spotting = any bloody vaginal discharge that required no sanitary pads or tampons per day. NOTE: Due to early termination of this study, the ENG-E2 reporting group received only up to 10 cycles of treatment, and the LNG-EE reporting group received only up to 9 cycles of treatment.
Time Frame: Up to 1 year
Population: FAS Evaluable population, defined as a subset of FAS population that met the following criteria: a) No more than 2 consecutive days with missing bleeding data on Daily Diary unless there was at least one day with BTB-S during the ring-use interval; and b) treatment cycle length (including hormone-free interval) is between 22 and 35 days, inclusive.
Measure: Count of Participants; unit: Participants
Arm/Group | ENG-E2 125 μg/300 μg | LNG-EE 150 μg/30 μg
Number analyzed (Participants) | 1504 | 492
Participants
  Cycle 2: number analyzed (Participants) | 1263 | 375
  Cycle 2 | 166 | 54
  Cycle 3: number analyzed (Participants) | 1001 | 295
  Cycle 3 | 112 | 36
  Cycle 4: number analyzed (Participants) | 755 | 231
  Cycle 4 | 79 | 20
  Cycle 5: number analyzed (Participants) | 483 | 155
  Cycle 5 | 42 | 13
  Cycle 6: number analyzed (Participants) | 295 | 88
  Cycle 6 | 29 | 8
  Cycle 7: number analyzed (Participants) | 125 | 40
  Cycle 7 | 13 | 7
  Cycle 8: number analyzed (Participants) | 36 | 10
  Cycle 8 | 8 | 2
  Cycle 9: number analyzed (Participants) | 7 | 1
  Cycle 9 | 1 | 0

5. Secondary Outcome: Number of Participants With Absence of Withdrawal Bleeding (AWB), by Cycle
Description: Participants were asked to keep a daily diary to record vaginal bleeding events. AWB was defined as no bleeding/spotting during the expected bleeding period. NOTE: Due to early termination of this study, the ENG-E2 reporting group received only up to 10 cycles of treatment, and the LNG-EE reporting group received only up to 9 cycles of treatment.
Time Frame: Up to 1 year
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | ENG-E2 125 μg/300 μg | LNG-EE 150 μg/30 μg
Number analyzed (Participants) | 1504 | 492
Participants
  Cycle 1: number analyzed (Participants) | 1448 | 441
  Cycle 1 | 76 | 15
  Cycle 2: number analyzed (Participants) | 1263 | 375
  Cycle 2 | 34 | 10
  Cycle 3: number analyzed (Participants) | 1001 | 295
  Cycle 3 | 26 | 10
  Cycle 4: number analyzed (Participants) | 755 | 231
  Cycle 4 | 17 | 6
  Cycle 5: number analyzed (Participants) | 483 | 155
  Cycle 5 | 3 | 0
  Cycle 6: number analyzed (Participants) | 295 | 88
  Cycle 6 | 3 | 1
  Cycle 7: number analyzed (Participants) | 125 | 40
  Cycle 7 | 0 | 2
  Cycle 8: number analyzed (Participants) | 36 | 10
  Cycle 8 | 0 | 1
  Cycle 9: number analyzed (Participants) | 7 | 1
  Cycle 9 | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to 1 year
Description: Safety analysis was based on all randomized participants in whom at least 1 vaginal ring was inserted or one comparator tablet was ingested. NOTE: Due to early termination of this study, the ENG-E2 reporting group received only up to 10 cycles of treatment, and the LNG-EE reporting group received only up to 9 cycles of treatment.
Arm/Group | ENG-E2 125 μg/300 μg | LNG-EE 150 μg/30 μg
Serious Adverse Events (participants affected / at risk) | 8/1504 | 3/492
Other Adverse Events (participants affected / at risk) | 116/1504 | 40/492
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ENG-E2 125 μg/300 μg (N=1504) | LNG-EE 150 μg/30 μg (N=492)
Visual acuity reduced (Eye disorders) | 0 (0) | 1 (1)
Dengue fever (Infections and infestations) | 1 (1) | 0 (0)
Gastrointestinal infection (Infections and infestations) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Foreign body (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Epilepsy (Nervous system disorders) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0)
Device deployment issue (Product Issues) | 1 (1) | 0 (0)
Cystitis haemorrhagic (Renal and urinary disorders) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ENG-E2 125 μg/300 μg (N=1504) | LNG-EE 150 μg/30 μg (N=492)
Headache (Nervous system disorders) | 116 (180) | 40 (68)

LIMITATIONS AND CAVEATS:
Because the trial was terminated early, participant diary data used for efficacy analysis and bleeding analysis were not verified. These results should be interpreted with caution. No hypothesis testing was performed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review all proposed abstracts, manuscripts or presentations regarding this trial 45 days prior to submission for publication/presentation. Any information identified by the Sponsor as confidential must be deleted prior to submission; this confidentiality does not include efficacy and safety results.